CLINICAL TRIAL: NCT06302348
Title: A Phase 3b Open-Label Study of Long-Term Neurocognitive Outcomes in Children With Phenylketonuria Treated With Sepiapterin
Brief Title: A Study of Sepiapterin in Participants With Phenylketonuria (PKU)
Acronym: EPIPHENY
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC923-PKU-401; 2024-514435-20-00 (Other: EU CT Number)
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Phenylketonuria
MeSH Terms: conditions — Phenylketonurias | interventions — sepiapterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sepiapterin (Experimental): Participants will receive age- and weight-adjusted doses of sepiapterin orally once daily for up to 6 years.
  Interventions: Drug: Sepiapterin

INTERVENTIONS:
Drug: Sepiapterin — Sepiapterin powder for oral use will be suspended in water or apple juice prior to administration.
  Other Names: PTC923; Sephience

SUMMARY:
The main purpose of this trial is to evaluate the long-term efficacy of sepiapterin on preserving neurocognitive functioning in children with PKU when treatment is initiated in early childhood.

DETAILED DESCRIPTION:
The study includes 2 parts: Part 1 and 2. Part 1 is an open-label sepiapterin-responsiveness test, and Part 2 is an open-label treatment period.

ELIGIBILITY:
Key Inclusion Criteria:

For all participants:

* Women of childbearing potential must have a negative pregnancy test at screening and agree to abstinence or the use of at least one highly effective form of contraception for the duration of the study, and for at least 90 days after the last dose of the study drug.
* Willing to maintain prescribed daily protein/Phe during Screening and Part 1.
* Established diagnosis of PKU with hyperphenylalaninemia (HPA) evidenced by at least 2 blood Phe measurement ≥600 micromoles (μmol)/liter (L) as documented in the medical history.
* For participants ≥1 month of age at Screening: A minimum of 1 documented blood Phe measurement <480 μmol/L within 1 month prior to Screening.
* For participants ≥1 month of age at Screening: Two screening blood Phe concentration values must be in the range ≥120 to ≤480 μmol/L.

For participants <1 month of age at the time of informed consent/assent only:

* Blood Phe at newborn screening ≥600 μmol/L.

For participants ≥30 months to <10 years of age:

* Baseline FSIQ score ≥80.

Key Exclusion Criteria:

* History of allergies or adverse reactions to any of the ingredients or excipients of synthetic tetrahydrobiopterin (BH4) or sepiapterin.
* Serious neuropsychiatric illness (for example, major depression) not currently under medical control or other concurrent disease or condition that, in the opinion of the investigator or sponsor, would interfere with the participant's ability to participate in the study or increase the risk of participation for that participant.
* Treatment with BH4 supplementation (sapropterin, KUVAN®) within 3 months prior to Screening.
* Current participation in another investigational drug study or use of any investigational agent within 30 days prior to Screening.
* Confirmed diagnosis of a primary BH4 deficiency as evidenced by biallelic pathogenic mutations in 6-pyruvoyltetrahydropterin synthase, recessive Guanosine-5'-triphosphate (GTP) cyclohydrolase I, sepiapterin reductase, quinoid dihydropteridine reductase, or pterin 4-alphacarbinolamine dehydratase genes.
* Any clinically significant laboratory abnormality as determined by the investigator.
* Any past medical history of an abnormal physical examination and/or laboratory findings indicative of signs or symptoms of renal disease, including calculated (Bedside Schwartz Equation) glomerular filtration rate (GFR) <60 milliliters (mL)/minute (min)/1.73 square meter (m^2).
* Major surgery within 90 days prior to Screening visit.

Note: Other protocol-defined inclusion and exclusion criteria may apply.

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2031-02-28 (Estimated); Study Completion 2031-02-28 (Estimated)

PRIMARY OUTCOMES:
Mean Change From Baseline in Full-scale Intelligence Quotient (FSIQ) Wechsler Preschool and Primary Scale of Intelligence - Fourth Edition (WPPSI-IV) Score | Baseline, Year 2
  Analysis for participants ≥30 months to <6 years of age.
Mean Change From Baseline in FSIQ Wechsler Intelligence Scale for Children - Fifth Edition (WISC-V) Score | Baseline, Year 2
  Analysis for participants ≥6 years to 16 years of age.

SECONDARY OUTCOMES:
Change From Baseline in Phenylketonuria-Quality of Life (PKU-QOL) Questionnaire Score | Baseline up to 4 years
Change From Baseline in the European Quality of Life - 5 Dimensions (EQ-5D) Score | Baseline up to 4 years
Mean Change From Baseline in FSIQ (WPPSI-IV) Score | Baseline, Year 4
  Analysis for participants aged ≥30 months to <6 years.
Mean Change From Baseline in FSIQ (WISC-V) Score | Baseline, Year 4
  Analysis for participants aged ≥6 years to 16 years.
Change From Baseline in Mean Blood Phenylalanine (Phe) Levels | Baseline up to 6 years

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University, Indianapolis, Indiana, United States